CLINICAL TRIAL: NCT05866848
Title: Effects of Caffeine on Cerebral Blood Flow in Clinically Healthy Young People
Brief Title: Effects of Caffeine on Cerebral Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde de Coimbra (Other)
Responsible Party: Principal Investigator, Helder Santos, PhD, Professor, Escola Superior de Tecnologia da Saúde de Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CCBF
Record Dates: First submitted 2023-04-06; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Cardiovascular System
Keywords: Transcranial Doppler ultrasonography; Middle Cerebral Artery; functional tests; cognitive activities; caffeine

STUDY DESIGN:
Intervention Model Description: All subjects were submitted to 2 evaluation moments: the first baseline moment and the second moment, 30 minutes after caffeine ingestion, which constitutes the time required for caffeine absorption.
  In each of the 2 moments, they performed 30 seconds of continuous breathing (hypoventilation), followed by 30 seconds of continuous rapid breathing (hyperventilation). VMCA measurements were stabilized between these tests. The study started with apnea testing because VMCA requires less time to return to baseline levels after hypoventilation than after hyperventilation.
  When VMCA measurements were stable, a 30-second baseline period was followed by three 30-second cognitive tasks, with a 1-minute break between activities: short-term memory test; solve a vocabulary problem; and solving a math problem. Three versions of each cognitive task were used for the three conditions. The procedure was completed with a final rest period of 60 seconds.
Who Masked: Participant
Masking Description: Three groups were randomly constituted, with 15 young people each: control group without caffeine, group with relatively small amount of caffeine (45 mg) administered and group with greater amount of caffeine (120 mg). Participants were not aware to which group they belong.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No caffeine (Placebo Comparator): The control group took flour capsules.
  Interventions: Other: Placebo
- Low caffeine (Experimental): Group with relatively small amount of caffeine (45 mg) administered.
  Interventions: Other: Anhydrous caffeine (45mg)
- High caffeine (Experimental): Group with greater amount of caffeine (120 mg) administered.
  Interventions: Other: Anhydrous caffeine (120mg)

INTERVENTIONS:
Other: Placebo — Flour capsules as a placebo.
  Arms: No caffeine
Other: Anhydrous caffeine (45mg) — Capsules dosed with 45mg of anhydrous caffeine.
  Arms: Low caffeine
Other: Anhydrous caffeine (120mg) — Capsules dosed with 120mg of anhydrous caffeine.
  Arms: High caffeine

SUMMARY:
The goal of this clinical trial is to evaluate in clinically healthy young people if:

* after caffeine ingestion, there are variations in blood velocity of the middle cerebral arteries (VMCA),
* this variation is dependent on the administered dose.

Transcranial Doppler ultrasonography was used to record blood VMCA in three groups of 15 clinically healthy young adults each - no caffeine, low caffeine (45 mg) and high caffeine group (120 mg). Transcranial Doppler ultrasonography provided simultaneous bilateral VMCA measurements while subjects performed functional tests (hyperventilation and hypoventilation orders) and three cognitive activities (Test 1, short-term remembering, Test 2, solving a vocabulary problem, and Test 3, solving a math problem) each in 31-second tests with 1-minute rest between them. Participants were assessed before and 30 minutes after caffeine ingestion.

DETAILED DESCRIPTION:
Were used in the study, Capsules dosed with 45mg and 120 mg of anhydrous caffeine and flour capsules as a placebo. In the preparation of the capsules, a semi-automatic capsulator No. 0 (Capsunorm® by Tecnyfarma®) were used, colorless hard gelatin capsules No. 0 by Acopharma® and anhydrous caffeine (Biochem®, C.A.S. 58-08-2).

Viasys Sonara transcranial Doppler unit and a 2 MHz probe were used to sample the middle cerebral artery at depths of 60 millimeters, using emission doppler pulsed performing spectral analysis in real time. Two probes (bilaterally) of 2MHz were placed at a depth between 55 and 60 mm, thus making it possible to analyse both middle cerebral arteries simultaneously.

Each participant was asked not to ingest caffeine and exercise vigorously for at least 12 hours before the assessment. In the case of smokers, they were also asked not to smoke for at least 2 hours before the evaluation. The laboratory had medium luminosity, silent and controlled temperature (23º/24ºC). To avoid inter-observer errors, all examinations were performed by the same investigator who was not aware of what dose was/had been administered to the participant.

Subjects were tested while seated in a reclining chair located in a dimly lit, sound-attenuated room and performed the activities with their eyes closed.

ELIGIBILITY:
Inclusion Criteria:

* clinically healthy young people

Exclusion Criteria:

* Individuals with hypertension, high cholesterol, diabetes, arrhythmias, carotid sinus syndrome, severe carotid stenosis and who were in an unstable clinical situation.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in Mean Velocity (Basal) | 30 minutes
  Changes in Mean Velocity, measure in m/s from baseline to 30 minutes after caffeine ingestion.
Changes in Mean Velocity (Hypoventilation) | 30 minutes
  By performing Hypoventilation, changes in Mean Velocity, measure in m/s from baseline to 30 minutes after caffeine ingestion.
Changes in Mean Velocity (Hyperventilation) | 30 minutes
  By performing Hyperventilation, changes in Mean Velocity, measure in m/s from baseline to 30 minutes after caffeine ingestion.
Changes in Mean Velocity (Short-term memory test) | 30 minutes
  With short-term memory test, changes in Mean Velocity, measure in m/s from baseline to 30 minutes after caffeine ingestion.
Changes in Mean Velocity (Vocabulary problem) | 30 minutes
  With solving vocabulary problems, changes in Mean Velocity, measure in m/s from baseline to 30 minutes after caffeine ingestion.
Changes in Mean Velocity (Math problem.) | 30 minutes
  With solving math problems, changes in Mean Velocity, measure in m/s from baseline to 30 minutes after caffeine ingestion.
Changes in Peak systolic velocity (Basal) | 30 minutes
  Changes in Mean Velocity, measure in m/s from baseline to 30 minutes after caffeine ingestion.
Changes in Peak systolic velocity (Hypoventilation) | 30 minutes
  By performing Hypoventilation, changes in Peak systolic velocity, measure in m/s from baseline to 30 minutes after caffeine ingestion.
Changes in Peak systolic velocity (Hyperventilation) | 30 minutes
  By performing Hyperventilation, changes in Peak systolic velocity, measure in m/s from baseline to 30 minutes after caffeine ingestion.
Changes in Peak systolic velocity (Short-term memory test) | 30 minutes
  With short-term memory test, changes in Peak systolic velocity, measure in m/s from baseline to 30 minutes after caffeine ingestion.
Changes in Peak systolic velocity (Vocabulary problems) | 30 minutes
  With solving vocabulary problems, changes in Peak systolic velocity, measure in m/s from baseline to 30 minutes after caffeine ingestion.
Changes in Peak systolic velocity (Math problems) | 30 minutes
  With solving math problems, changes in Peak systolic velocity, measure in m/s from baseline to 30 minutes after caffeine ingestion.
Changes in Vend-diastolic velocity (Basal) | 30 minutes
  Changes in Mean Velocity, measure in m/s from baseline to 30 minutes after caffeine ingestion.
Changes in Vend-diastolic velocity (Hypoventilation) | 30 minutes
  By performing Hypoventilation, changes in Vend-diastolic velocity, measure in m/s from baseline to 30 minutes after caffeine ingestion.
Changes in Vend-diastolic velocity (Hyperventilation) | 30 minutes
  By performing Hyperventilation, changes in Vend-diastolic velocity, measure in m/s from baseline to 30 minutes after caffeine ingestion.
Changes in Vend-diastolic velocity (Short-term memory test) | 30 minutes
  With short-term memory test, changes in Vend-diastolic velocity, measure in m/s from baseline to 30 minutes after caffeine ingestion.
Changes in Vend-diastolic velocity (Vocabulary problems) | 30 minutes
  With solving vocabulary problems, changes in Vend-diastolic velocity, measure in m/s from baseline to 30 minutes after caffeine ingestion.
Changes in Vend-diastolic velocity (Math problems) | 30 minutes
  With solving math problems, changes in Vend-diastolic velocity, measure in m/s from baseline to 30 minutes after caffeine ingestion.

SECONDARY OUTCOMES:
Changes in Heart Rate (Basal) | 30 minutes
  Changes in Heart Rate, measure in bpm from baseline to 30 minutes after caffeine ingestion.
Changes in Heart Rate (Hypoventilation) | 30 minutes
  By performing Hypoventilation, changes in Heart Rate, measure in bpm from baseline to 30 minutes after caffeine ingestion.
Changes in Heart Rate (Hyperventilation) | 30 minutes
  By performing Hyperventilation, changes in Heart Rate, measure in bpm from baseline to 30 minutes after caffeine ingestion.
Changes in Heart Rate (Short-term memory test) | 30 minutes
  With short-term memory test, changes in Heart Rate, measure in bpm from baseline to 30 minutes after caffeine ingestion.
Changes in Heart Rate (Vocabulary problems) | 30 minutes
  With solving vocabulary problems, changes in Heart Rate, measure in bpm from baseline to 30 minutes after caffeine ingestion.
Changes in Heart Rate (Math problems) | 30 minutes
  With solving math problems, changes in Heart Rate, measure in bpm from baseline to 30 minutes after caffeine ingestion.

CONTACTS AND LOCATIONS:
Overall Officials: Hélder Santos, PhD, Principal Investigator — Polytechnic Institute of Coimbra - Coimbra Health School
Locations (1):
- Coimbra Health School, Coimbra, Portugal

REFERENCES:
- [Derived] Gaspar C, Rocha C, Balteiro J, Santos H. Effects of caffeine on cerebral blood flow. Nutrition. 2024 Jan;117:112217. doi: 10.1016/j.nut.2023.112217. Epub 2023 Sep 6. PMID 37826937